CLINICAL TRIAL: NCT05523999
Title: Evaluation of the Optimal Time of Recognition of a Cardiac Arrest Within the EMS 95
Brief Title: Recognition of a Cardiac Arrest Within the EMS
Acronym: ACR90
Status: Recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD2321
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Arrest
Keywords: cardiorespiratory arrest (CRA); Medical Regulation Assistant (MRA); EMS; External Cardiac Massage; External Automated Defibrillator; 90 seconds
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Time elapsed between the taking in charge of the call and the recognition of a cardiac arrest by the MRA — Prospective study within the EMS 95, to evaluate if the maximum delay of 90 seconds between the call to the EMS and the recognition of the cardiac arrest is reached.

SUMMARY:
This study aims to evaluate the average time taken by the Medical Regulation Assistants (MRA) to detect a cardiac arrest during the call to the EMS as well as the factors influencing this delay.

Its main objective is to evaluate the delay, in seconds, between the call being picked up and the recognition of a cardiac arrest by the medical regulation assistant at the EMS 95

DETAILED DESCRIPTION:
In France, the incidence of cardiac arrest in adults is approximately 40,000 per year. It is a major cause of mortality with an average survival rate of 8%, as well as morbidity, particularly neurological morbidity for surviving patients. The majority of cardiac arrests occur at In France, the incidence of cardiac arrest in adults is approximately 40,000 per year. It is a major cause of mortality with an average survival rate of 8%, as well as morbidity, particularly neurological morbidity for surviving patients. The majority of cardiac arrests occur at home, in the presence of a witness.

In the event of a cardiac arrest, every minute counts. Studies have shown that the time between the patient's collapse and the start of ECM (External Cardiac Massage) is directly correlated to the survival rate after a cardiac arrest.

According to other studies, a maximum delay of 90 seconds between the call to the EMS and the recognition of the cardiac arrest would be the most optimal for the patient, but is it reached at the EMS 95? This study aims at evaluating the average time taken by the Assistants of Medical Regulation (ARM) to detect a cardiac arrest during the call to the EMS as well as the factors influencing this delay.

Its main objective is to evaluate the delay, in seconds, between the call pick-up and the recognition of a cardiac arrest by the medical regulation assistant at the EMS 95. This evaluation will be made in particular by determining the elements of language highlighting the cardiac arrest, those which lengthen the time of detection of the arrest and the delay of starting a procedure by the ARM. The study will be conducted within the EMS and will include a review of the current state of knowledge and experience of the MRAs. This study will be carried out within the EMS 95.

ELIGIBILITY:
Inclusion Criteria :

- Any call resulting in the detection of a cardiac arrest during ARM regulation: calls to 15 and calls transmitted by 18

Exclusion Criteria :

* Traumatic context
* Call involving cardiac arrest already identified as such by the caller or 18
* Call with criteria of proven death
* The caller does not speak French, the linguistic elements noted are not usable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical regulation assistant taking a call from a witness of a cardiac arrest between 01/01/2024 and 30t/04/2024
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation, of the time elapsed (seconds) between the taking in charge of the call and the recognition of a cardiac arrest by the medical regulation assistant (ARM) of the EMS 95. | At the end of the study, an average of 5 month
  Measure of the time in seconds between picking up the phone and the recognition of the cardiac arrest by the medical regulation assistant

SECONDARY OUTCOMES:
Identify language that highlights cardiac arrest | At the end of the study, an average of 5 month
  Collection of the initial reason for appeal and everything said by the witness that may point to cardiac arrest
Identify language that increases the time to detect cardiac arrest | At the end of the study, an average of 5 month
  Collection of everything said by the witness increasing the detection of the cardiac arrest
Evaluation of the time required for the MRA to initiate a procedure (AED search: External Automated Defibrillator or initiation of external cardiac massage assistance) | At the end of the study, an average of 5 month
  Collection of time (seconds) between :
  * the MRA taking the call and requesting an AED search
  * the MRA taking the call and the start of external cardiac massage
Identification of factors that may influence the time to recognition of cardiac arrest (MRA experience, tone of the call) | At the end of the study, an average of 5 month
  Collection of call tone (witness anxiety level) and MRA experience in years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ariane Zoya-Gillet, Principal Investigator — Hôpital NOVO
Locations (1):
- EMS department - Hospital René Dubos - Pontoise, Pontoise, France

IPD SHARING:
Plan to Share IPD: No